CLINICAL TRIAL: NCT06666946
Title: Efficacy and Safety Study of Early Electroacupuncture Treatment Combined With ICU Standard Therapy on Organ Dysfunction and Clinical Outcomes in Patients With Sepsis: a Single-center, Randomized, Sham-Controlled Trial
Brief Title: Efficacy and Safety of Electroacupuncture for ICU Sepsis Patients
Acronym: SEPSIS-ACU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shusheng Li (Other)
Responsible Party: Sponsor-Investigator, Shusheng Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEPSIS-ACU(20240730); 2022YFC3500704 (Other Grant/Funding Number: The National Key Research and Development Program)
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-10

CONDITIONS: Sepsis
Keywords: sepsis; electroacupuncture; organ dysfunction; inflammation; immune
MeSH Terms: conditions — Sepsis; Inflammation | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EA group (Experimental): For the EA group, participants will be assigned to receive 6 sessions of EA applied at bilateral acupoints Zusanli (ST36) and Yanglingquan (GB34), once daily, with the first session of EA applied within 24 hours after randomization.
  Interventions: Device: Electroacupuncture
- Sham EA group (Sham Comparator): For the sham EA group, participants will be assigned to receive 6 sessions of sham EA on two sham points, once daily, with the first session of sham EA applied within 24 hours after randomization.
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Hwato brand disposable acupuncture needles (size 0.30 × 40 mm), and SDZ-V EA apparatuses will be used. Participants in the EA group will receive acupuncture at bilateral ST36 and GB34. After sterilisation, sterile adhesive pads will be placed on bilateral ST36 and GB34, and acupuncture needles will be inserted through the adhesive pads approximately 20 to 30 mm into the skin. Following needle insertion, manual manipulation of needles will be performed on all needles to reach de qi (a composite of sensations including soreness, numbness, distention, heaviness, and other sensations). Then, paired electrodes from the EA apparatus will be attached transversely to the needle handles at bilateral ST36 and GB34. EA stimulation lasted for 30 minutes with a continuous wave of 10 Hz and a current intensity of 0.5 to 1 mA (preferably with the skin around the acupoints shivering mildly without pain). Participants will receive 6 treatment sessions once daily for 6 consecutive days.
  Arms: EA group
Device: Sham electroacupuncture — Non-insertive placebo needles (size 0.30 × 30 mm), and SDZ-V EA apparatuses will be used. Participants in the sham EA group will receive sham EA with a non-insertive placebo needle on sham acupoints. The sham ST36 point is located at 1 cun (≈20 mm) lateral to ST36, and the sham GB34 point is located at 1 cun (≈20mm) lateral to GB 34. Procedures, electrode placements, and other treatment settings will be the same as in the EA group but with no skin penetration, electricity output, or de qi.
  Arms: Sham EA group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of electroacupuncture (EA) combined with standard Intensive Care Unit (ICU) therapy on organ dysfunction and other clinical outcomes in sepsis patients. Additionally, this study will conduct subgroup analyses to investigate the influence of septic shock and immunomodulators on the treatment effects and their correlation with electroacupuncture efficacy.

DETAILED DESCRIPTION:
The proposed single-center, participant-blind, two arms, randomized, sham-controlled clinical trial is to evaluate the efficacy and safety of electroacupuncture (EA) combined with standard Intensive Care Unit (ICU) therapy on organ dysfunction and other clinical outcomes in sepsis patients. We planned to conduct this single-center trial in Tongji Hospital, affiliated to Huazhong University of Science and Technology (HUST). Patients, who are initially diagnosed with sepsis, will be assessed for eligibility within 24 hours of their ICU admission. Then, eligible participants will be informed and randomly assigned to one of the two groups: the EA group or the sham EA group, in a 1:1 ratio using block randomization. Patients will receive the first EA/sham EA therapy within 24 hours after randomization. The treatment will be administered once daily for 6 days continuously, and followed by 28 days after randomization. The primary outcome will be the SOFA score at Day 7 after randomization. Secondary outcomes include mortality, ICU-free days, hospital-free days, organ-support-free days at Day 28. SOFA score components and related serological results will also be included. Data collection will be conducted by an electronic data management system. Data analyses will be performed on a full analysis set and a per protocol set.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, and gender is not limited.
* 2. Meets the diagnostic criteria of Sepsis (Sepsis-3): In patients with infection or suspected infection, Sepsis is diagnosed when the Sequential (Sepsis related) Organ Failure Assessment (SOFA) score increased by ≥2 points from baseline.
* 3. Patients or their legal representatives understand and voluntarily sign the informed consent for this study.

Exclusion Criteria:

* 1. Patients with lower extremity denervation.
* 2. Patients with lower extremity amputation or congenital disability with lower limb hypoplasia.
* 3. Patients with severe acute trauma such as active bleeding or unfixed fractures in the lower extremities.
* 4. Patients with skin damage, infection, bleeding, or hematoma near the lower extremity acupuncture site.
* 5. Patients with implantable medical devices, such as pacemakers, implantable cardioverter defibrillators (ICD) or deep brain stimulation (DBS).
* 6. Patients who are pregnant, breast feeding during the study.
* 7. Patients whose expected duration of ICU length of stay is less than 48 hours.
* 8. Patients whose legal representatives refuse routine active treatment and sign palliative treatment consent.
* 9. Patients who are currently participating in another randomized clinical trial.
* 10. Patients or their legal representatives refused to participate in the study or were unable to sign informed consent.
* 11. Immunosuppressive status, including but not limited to: congenital immunosuppressive patients, AIDS patients, organ transplant patients, long-term use of immunosuppressive patients, patients receiving tumor radiotherapy or chemotherapy within 1 month;
* 12. Patients with an anticipated survival prognosis of no more than 7 days due to advanced disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the SOFA score between baseline and 7 days after randomization | At baseline (before randomization), and every day after the first treatment to day 7 after randomization
  The SOFA (Sequential Organ Failure Assessment) score was based on six different scores, one for each of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems each scored from 0 to 4 with an increasing score reflecting worsening organ dysfunction.

SECONDARY OUTCOMES:
All-cause mortality at day 28 | At day 28 after randomization
  It refers to the total number of patients who die from any cause within 28 days of being admitted to the hospital. It will be described as a ratio.
All-cause ICU mortality at day 28 | At day 28 after randomization
  It refers to the total number of patients who die in the ICU from any cause within 28 days of being admitted to the hospital. It will be described as a ratio.
ICU-free days to day 28 | At day 28 after randomization
  The number of days from the patient's discharge from the ICU to the 28th day after randomization is calculated. If the patient re-enters the ICU, the total number of days without ICU care is subtracted from the number of days spent in the ICU.
Hospital-free days to day 28 | At day 28 after randomization
  The number of days from the patient's discharge to the 28th day after randomization is calculated. If the patient re-enters the hospital, the total number of days without hospital care is subtracted from the number of days spent in the hospital.
Ventilator-free time to day 28 | At day 28 after randomization
  This refers to the period from randomization to the 28th day, during which the patient must be alive and have at least 48 hours off the ventilator. Subtract the time that the ventilator was required again from the total time. If the patient dies in the hospital after being off the ventilator, the value is set to 0.
Vasopressor-free days to day 28 | At day 28 after randomization
  From randomization to the 28th day, this refers to the time the patient is alive and has not received vasopressor medications for at least 4 hours. If the patient dies in the hospital after discontinuing the medication, the value is set to 0.
CRRT-free days to day 28 | At day 28 after randomization
  The time from randomization to the 28th day during which the patient did not use continuous renal replacement therapy(CRRT).
SOFA score at Day 8 and 9 after randomization | At day 8 and 9 after randomization
  After-effect assessed by SOFA score, which is same as the description of the primary outcome.
SOFA score of each system | At baseline (before randomization), and every day after the first treatment to day 9 after randomization
  Independent scores for each system that makes up the SOFA score
SOFA score components | At baseline (before randomization), and every day after the first treatment to day 9 after randomization
  ie, PaO2 to FiO2 ratio, ventilator use, platelet counts, total bilirubin, MAP, vasopressor use, creatinine level, urine volume
Liquid equilibrium parameter | At baseline (before randomization), and every day after the first treatment to day 6 after randomization
  Daily fluid intake, output and fluid balance of ICU patients will be recorded continuously.

OTHER OUTCOMES:
Serum biomarkers and related cellular assays | At baseline (before randomization), day 3 and day 7
  TNF-α, IL-6 , IL-1β, IL-8, IL-4 and IL-10 in pg/ml; C-reactive protein (CRP) in mg/L; Procalcitonin (PCT) in ng/ml; Serum soluble programmed cell death protein (sPD-1) levels in pg/ml; Acetylcholine (ACh) in μmol/L; Choline acetyltransferase (ChAT) in μg/L; CD3+ cell fraction, CD4+ cell fraction, CD3+/CD4+ T cell ratio, percentage of NK cells to total lymphocytes, and ratio of neutrophils to lymphocytes (N/L) in percentage.
Adverse events related to EA or sham EA | From the beginning of acupuncture , up to 1 hour after the end of each 30 min duration of acupuncture.
  Outcome assessors will record adverse events after each treatment, including bleeding, subcutaneous haemorrhage, serious pain, and local infection.

CONTACTS AND LOCATIONS:
Overall Officials: Shusheng Li, PhD., Principal Investigator — Tongji Hospital
Locations (1):
- Department of Critical Care Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
IPD after de-identification can be shared on individual request to the principal investigator at lishusheng@hust.edu.cn.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available for two years after the publication of the primary outcomes.